CLINICAL TRIAL: NCT06059313
Title: Relationship Between Premorbid Personality Traits and Cognitive and Behavioral Disorders
Brief Title: Premorbid Personality Profile of Patients With Cognitive and Behavioral Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0343
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Behavioral Variant of Frontotemporal Disorder (bvFTD); Phenocopy Frontotemporal Dementia (phFTD); Frontal Variant of Alzheimer Disease; Bipolar Disorder
Keywords: bvFTD; fvAD; phFTD; bipolar disorder,personality
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Behavioral variant of frontotemporal disorder (bvFTD): A group of participants who fulfill Rascovsky criteria (2011) for behavioural variant Frontotemporal Dementia
  Interventions: Other: Submission of the NEO-PI-3 questionnaire; Other: Submission of the Interpersonal Reactivity Index questionnaire (IRI)
- Phenocopy frontotemporal dementia (phFTD): A group of participants who fulfill who fulfill Rascovsky criteria (2011) for possible behavioural variant Frontotemporal Dementia and have no imaging abnormalities.
  Interventions: Other: Submission of the NEO-PI-3 questionnaire; Other: Submission of the Interpersonal Reactivity Index questionnaire (IRI)
- Frontal variant of Alzheimer disease: A group of participants who fulfill Ossenkopele criteria (2022)
  Interventions: Other: Submission of the NEO-PI-3 questionnaire; Other: Submission of the Interpersonal Reactivity Index questionnaire (IRI)
- Bipolar disorder: A group of participants who fulfill CIM 10 criteria
  Interventions: Other: Submission of the NEO-PI-3 questionnaire; Other: Submission of the Interpersonal Reactivity Index questionnaire (IRI)

INTERVENTIONS:
Other: Submission of the NEO-PI-3 questionnaire — The questionnaire contains 240 statements. For each statement, the patient chooses the answer that best corresponds to their choice (FD: strongly disagree - D: disagree - N: neutral - A: agree - FA: strongly agree).
Other: Submission of the Interpersonal Reactivity Index questionnaire (IRI) — The test assesses two cognitive and two affective components of empathy that influence each other and affect attitudes and behaviors toward others.

SUMMARY:
Damages in frontal area present in neurodegenerative disease (frontotemporal degeneration, frontal variant of Alzheimer disease) and in psychiatric disease (bipolar disorder) can affect behavior and cognition including social cognition. Symptoms vary both quantitatively and qualitatively from disease to another and from person to person. It cannot be completely excluded that in some cases, factors of susceptibility such as premorbid personality traits lead to frontal fragility.

The study will assess the relationship between premorbid profile using NEO-PI 3 inventory and cognitive and behavioral/psychobehavioral manifestations in patients with behavioral variant of frontotemporal disorder (bvFTD), phenocopy frontotemporal dementia (phFTD), frontal variant of Alzheimer disease, bipolar disorder characterized with frontal damages.

ELIGIBILITY:
Inclusion Criteria :

* Patients with behavioral variant of frontotemporal disorder (bvFTD) according to Rascovsky criteria (2011) or patients with phénocopy frontotemporal dementia (phFTD) who fulfill criteria for possible bvFTD and have no imaging abnormalities or patients with frontal variant of Alzheimer disease according to Ossenkopele criteria (2022), or patient with bipolar disorder according to CIM 10 criteria
* Score for Mini-mental state examination ≥ 18
* Patient with caregiver who has who has known him/her in the 10 years preceding the disease onset.
* Patient and caregiver consents (no opposition)

Exclusion Criteria :

* Patient with no caregiver
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted among eligible patients with bvFTD, fvAD, phFTD, followed to Memory Resource and Research Centre at Nantes university Hospital CMRR or referred to the department for a neuropsychological assessment (bipolar disorder). It will prospectively enroll 120 participants.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Premorbid personality traits | Baseline
  Premorbid personality traits will be assessed by the NEO- NEO Personality Inventory-3 (NEO-PI-3). The NEO PI-3 measures the five major domains of personality: Neuroticism, Extraversion, Openness to experience, Conscientiousness and Agreeableness. Each domain is defined by 6 facets. NEOPI-3 includes 240 items and responses are made on a 5-point Likert -type scale ranging from strongly Disagree to strongly agree. The NEOPI 3 will be completed by a caregiver who has known the patient in the 10 years preceding the disease onset.

SECONDARY OUTCOMES:
Interpersonal Reactivity Index (IRI) | Baseline
  IRI is a 28-item questionnaire measuring 4 aspects of empathy : perspective-taking, fantasy, empathic concern, personal distress. Each answer is rated from 1 (does not describe me well) to 5 (describes me very well).

IPD SHARING:
Plan to Share IPD: No